CLINICAL TRIAL: NCT03254823
Title: Defining Autoimmune Aspects of Myalgic Encephalomyelitis/Chronic Fatigue Syndrome (ME/CFS)
Brief Title: Autoimmunity in Myalgic Encephalomyelitis/Chronic Fatigue Syndrome (ME/CFS)
Status: Completed | Type: Observational
Sponsor: University of East Anglia (Other)
Collaborators: Quadram Institute Bioscience (Other); Invest in ME Research UK (Unknown)
Responsible Party: Sponsor
Other Study IDs: 17/LO/1102
Record Dates: First submitted 2017-07-26; First posted 2017-08-21 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2022-10

CONDITIONS: Myalgic Encephalomyelitis; Chronic Fatigue Syndrome
MeSH Terms: conditions — Fatigue Syndrome, Chronic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Biospecimen Retention: Samples With DNA — faecal samples serum plasma peripheral blood mononuclear cells
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Severe ME/CFS patients: patients with a clinical diagnosis of ME/CFS and are house or bed bound.
- Household controls: Healthy human participants who are either related/non-related to, living in the same household or in close proximity to, or providing care to the severe ME/CFS patient they are paired with. They are used as an environmental control.

SUMMARY:
This study investigates whether there is an immune response directed against gut microbes or food and parts of the body in severe Myalgic Encephalomyelitis/Chronic Fatigue Syndrome (ME/CFS) patients.

DETAILED DESCRIPTION:
Severe Myalgic Encephalomyelitis/Chronic Fatigue Syndrome (ME/CFS) patients will be identified by Epsom and St Helier CFS Service and the Clinical Research Network Eastern. Information sheets will be posted by health professionals to eligible patients. Interested patients are asked to arrange a telephone call with the research team to receive more information about the study. Volunteers still interested after the 72 hour consideration period arrange a home visit to be taken through the consenting process.

Household controls will be recruited through patients participating in the study. Patients invited will be provided with information about household controls. The patient identifies and informs potential household controls of the study using information sheets provided by their health professional. Household controls willing to participate in the study will be taken through an eligibility questionnaire with GCP trained researchers.

Six stool and blood samples will be collected over the three year study period. Stool and blood samples need to be collected within 24 hours of each other, during home visits. 48 hour food diaries will be completed prior to each stool sample collection.

The study is based at the Quadram Institute and the University of East Anglia (UEA). The research is funded by the UEA and Invest in ME Research UK.

ELIGIBILITY:
Inclusion Criteria:

* severe ME/CFS patients: men or women aged 18 to 70 years with a clinical diagnosis of severe ME/CFS patients
* household controls: men or women aged 18 to 70 years, no current or on-going medical conditions. Has to be either related/non-related, living in the same household or in close proximity to, or providing care to the severe ME/CFS patient they are paired with.

Exclusion Criteria:

* severe ME/CFS patients: the presence of significant anxiety or depression. Have received probiotics or antibiotics up to six weeks before joining the study.
* Household controls: The presence of long term medical conditions, in particular, affecting the stomach or bowel. Previously diagnosed with autoimmune diseases, for example, systemic lupus erythematous or rheumatoid arthritis. Suffer from significant anxiety or depression. In recipient of immunomodulatory drugs, statins, beta blocker or steroids. Have received probiotics or antibiotics up to six weeks before joining the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Severe ME/CFS patient attending Epsom and St Helier CFS Clinic will be identified by the Director of the clinic, Dr Bansal. CRN Eastern will notify general practitioners and occupational therapists of the study. They will then identify severe ME/CFS patients in the East of England.
  Household controls will be recruited through severe ME/CFS patients participating in the study.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2017-08-09 (Actual); Primary Completion 2022-08-30 (Actual); Study Completion 2022-08-30 (Actual)

PRIMARY OUTCOMES:
Measurement of antibody levels | 3 years
  Measurement of serum antibodies that are reactive with intestinal microbes or foods. Antibody levels will reflect the presence of an immune response directed against gut microbes in severe ME/CFS patients.
Measurement of cellular immune responses | 3 years
  Measurement of memory T and memory B cells (from peripheral blood mononuclear cells in the blood) specific to gut microbes (from stool sample). The presence of memory T and B cells will indicate a systemic (whole body) immune response directed against gut microbes in severe ME/CFS patients.
Expression of microbial and viral DNA/RNA | 3 years
  To identify the bacterial, fungal and virus populations in stool samples.

SECONDARY OUTCOMES:
Measurement of autoimmunity | 3 years
  Measurement of serum antibodies and immune cells that are reactive with human cells, such as cells of the central nervous system. The presence of an immune response against human cells and human cell proteins is indicative of the presence of autoimmunity.

CONTACTS AND LOCATIONS:
Overall Officials: Simon Carding, Principal Investigator — Quadram Institute Bioscience
Locations (1):
- Quadram Institute, Norwich, United Kingdom

IPD SHARING:
Plan to Share IPD: No